CLINICAL TRIAL: NCT05590091
Title: Allogeneic Hematopoietic Stem Cell Transplantation Based on the Support of Intelligent Nutrition Management System Nutritional Intervention Research in Recipients During Peritransplantation
Brief Title: Study on Intelligent Nutrition Support Therapy for Hematopoietic Stem Cell Transplantation Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: DPJG-Y-202205
Record Dates: First submitted 2022-09-13; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Nutrition Aspect of Cancer; Stem Cell Transplant Complications
Keywords: HSCT; Nutrition therapy; Intestinal graft-versus-host disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): roup A were given precise dietary guidance and enteral and parenteral nutrition support treatment using only nutrition software. It is recommended that the precise recommended time covers the start of enrollment until 100 days after transplantation
  Interventions: Other: Parenteral nutrition;Enteral nutrition
- The control group (No Intervention): Group B patients were given the routine nutritional support treatment plan commonly used in clinics. Patients in both groups were monitored and followed up at -5d before transplantation and at +6d, +30d, +60d, +100d, +180d, and +360d after transplantation.

INTERVENTIONS:
Other: Parenteral nutrition;Enteral nutrition — The intelligent nutrition management system was used to carry out standardized nutrition management of patients after hematopoietic stem cell transplantation
  Arms: Experimental group

SUMMARY:
The use of high-dose radiotherapy, chemotherapy and preventive antibiotics in the preconditioning regimen before allogeneic hematopoietic stem cell transplantation can easily lead to damage to the gastrointestinal mucosa, resulting in malnutrition, and even progression to cachexia, which directly leads to multiple organ failure; The damage of the intestinal mucosal barrier, secondary to the translocation of intestinal-derived bacteria, leads to bloodstream infection and lung infection (drug-resistant Enterobacteriaceae, especially carbapenem-resistant Enterobacteriaceae infection) is one of the challenges faced in clinical treatment. A major problem that affects the long-term survival rate of patients. Nutrition therapy based on the support and guidance of the intelligent nutrition management system aims to improve the adherence and compliance rate of patients with nutritional support therapy through scientific and accurate monitoring and intervention, thereby improving the nutritional status of patients and improving the tolerance of patients to radiotherapy and chemotherapy， and reduce the incidence of adverse reactions. At the same time, it is expected that nutritional support therapy will protect the integrity of the intestinal mucosal barrier of patients, reduce the incidence of enterobacteriaceae bacterial infections (mainly drug-resistant Klebsiella pneumoniae and Escherichia coli infections), and ultimately improve the long-term survival rate. Purpose.

This trial objects are patients who are going to undergo allogeneic hematopoietic stem cell transplantation, and explores the use of intelligent nutrition management system for data support to reduce the incidence and severity of malnutrition, especially cachexia, and to help reduce the incidence and severity of Enterobacteriaceae bacterial infections. It can reduce the incidence of acute intestinal GVHD and ultimately improve the long-term survival rate and quality of life of patients.

DETAILED DESCRIPTION:
1. Background The use of high-dose radiotherapy, chemotherapy and preventive antibiotics in the preconditioning regimen before allogeneic hematopoietic stem cell transplantation can easily lead to damage to the gastrointestinal mucosa, resulting in malnutrition, and even progression to cachexia, which directly leads to multiple organ failure; The damage of the intestinal mucosal barrier, secondary to the translocation of intestinal-derived bacteria, leads to bloodstream infection and lung infection (drug-resistant Enterobacteriaceae, especially carbapenem-resistant Enterobacteriaceae infection) is one of the challenges faced in clinical treatment. A major problem that affects the long-term survival rate of patients. Nutrition therapy based on the support and guidance of the intelligent nutrition management system aims to improve the compliance and compliance rate of patients with nutritional support therapy through scientific and accurate monitoring and intervention, thereby improving the nutritional status of patients and improving the tolerance of patients to radiotherapy and chemotherapy. Reduce the incidence of adverse reactions. At the same time, it is hoped that nutritional support therapy will protect the integrity of the intestinal mucosal barrier of patients, reduce the incidence of Enterobacteriaceae bacterial infections (mainly drug-resistant Klebsiella pneumoniae and Escherichia coli infections), and ultimately improve the long-term survival rate.
2. Purposes To investigate the effect of continuous nutritional therapy on the nutritional status of allogeneic HSCT recipients based on an intelligent nutritional management system, and to reduce the incidence of malnutrition during peri-transplantation.
3. Conditions to be met to participate in a study/trial Inclusion criteria: 1. Age 12-55 years old; 2. Patients who are about to receive allo-HSCT (1-2 weeks before pretreatment) ; 3. No serious medical and surgical complications, no mental and psychological diseases; 4. . Those who voluntarily participate in the study and sign the informed consent in writing. 4. No serious allergic diseases, especially those with milk protein allergy; Exclusion criteria: 1. Physical discomfort during the test; 2. Complicated with severe infection or other serious underlying diseases, and the duration of hemodynamic instability is ≥5 days; 3. Severe liver and kidney dysfunction and coagulation disorders persist Time ≥ 5 days; 4. Intractable cachexia phase/refractory phase: tumor continues to progress, no response to treatment; catabolism is active, and body weight continues to lose weight that cannot be corrected 5. Being unable to understand or comply with the research protocol due to clinical symptoms of brain dysfunction or severe mental illness; 6. drug abuse, medical, psychological or social conditions that may interfere with the subject's participation in the research or the evaluation of the research results; 7. Those who cannot be followed up as scheduled; 8. The investigator believes that the subject has any clinical or laboratory abnormalities or compliance problems that are not suitable for participation in this clinical study.
4. Number of trail subjects This clinical trial is a randomized controlled trial, and plans to recruit a total of 106 subjects, with 53 subjects in the experimental group and 53 in the control group .
5. Research/Trial Process This study is a randomized controlled clinical trial. After signing the informed consent, the subjects who meet the inclusion and exclusion criteria will be randomly assigned to the experimental group and the control group at a ratio of 1:1. The control group only receives conventional treatment, while the experimental group receives precise nutritional intervention with the assistance of an intelligent nutrition system. The intervention period of the experimental group will be 100 days after being enrolled and receiving the transplantation. The patients in the control group and experimental group will be followed up at -5d before transplantation and +6d, +30d, +60d, +100d, +180d, and +360d after transplantation. .

Randomized trial : The grouping is randomly performed by the computer, so that the bias caused by the grouping can be avoided. Each subject had a 50% chance of being assigned to both the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-55 years old;
* Patients who are about to receive allo-HSCT (1-2 weeks before pretreatment);
* No serious medical and surgical complications, no mental and psychological diseases;
* Those who voluntarily participate in the research and sign the informed consent.
* No serious allergic diseases, especially those with milk protein allergy

Exclusion Criteria:

* Feeling unwell during the test;
* Combined with severe infection or other serious underlying diseases, the duration of hemodynamic instability is ≥5 days;
* Severe liver and kidney dysfunction and coagulation disorder for ≥5 days;
* Intractable cachexia/refractory stage: the tumor continues to progress and does not respond to treatment; the catabolism is active, and the body weight continues to lose weight that cannot be corrected
* Clinical symptoms of brain dysfunction or severe mental illness, unable to understand or comply with the research protocol;
* Drug abuse, medical, psychological or social conditions that may interfere with the subject's participation in the research or the evaluation of the research results;
* Those who cannot be followed up as scheduled;
* The investigator believes that the subjects have any clinical or laboratory abnormalities or compliance problems and are not suitable to participate in this clinical study

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who fell sick and vomit at certain checkpoint of transplantation | 5 days before transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of sick and vomit and statistics the number of participants who developed these symptoms
Number of participants who fell sick and vomit at certain checkpoint of transplantation | 6 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of sick and vomit and statistics the number of participants who developed these symptoms
Number of participants who fell sick and vomit at certain checkpoint of transplantation | 30 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of sick and vomit and statistics the number of participants who developed these symptoms
Number of participants who fell sick and vomit at certain checkpoint of transplantation | 60 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of sick and vomit and statistics the number of participants who developed these symptoms
Number of participants who fell sick and vomit at certain checkpoint of transplantation | 100 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of sick and vomit and statistics the number of participants who developed these symptoms
Number of participants who fell sick and vomit at certain checkpoint of transplantation | 180 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of sick and vomit and statistics the number of participants who developed these symptoms
Number of participants who fell sick and vomit at certain checkpoint of transplantation | 360 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of sick and vomit and statistics the number of participants who developed these symptoms
Number of participants who fell constipate at certain checkpoint of transplantation | 5 days before transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of constipate and statistics the number of participants who developed these symptoms
Number of participants who fell constipate at certain checkpoint of transplantation | 6 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of constipate and statistics the number of participants who developed these symptoms
Number of participants who fell constipate at certain checkpoint of transplantation | 30 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of constipate and statistics the number of participants who developed these symptoms
Number of participants who fell constipate at certain checkpoint of transplantation | 60 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of constipate and statistics the number of participants who developed these symptoms
Number of participants who fell constipate at certain checkpoint of transplantation | 100 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of constipate and statistics the number of participants who developed these symptoms
Number of participants who fell constipate at certain checkpoint of transplantation | 180 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of constipate and statistics the number of participants who developed these symptoms
Number of participants who fell constipate at certain checkpoint of transplantation | 360 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of constipate and statistics the number of participants who developed these symptoms
Number of participants who fell difficulty urinating at certain checkpoint of transplantation | 5 days before transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of difficulty urinating and statistics the number of participants who developed these symptoms
Number of participants who fell difficulty urinating at certain checkpoint of transplantation | 6 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of difficulty urinating and statistics the number of participants who developed these symptoms
Number of participants who fell difficulty urinating at certain checkpoint of transplantation | 30 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of difficulty urinating and statistics the number of participants who developed these symptoms
Number of participants who fell difficulty urinating at certain checkpoint of transplantation | 60 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of difficulty urinating and statistics the number of participants who developed these symptoms
Number of participants who fell difficulty urinating at certain checkpoint of transplantation | 100 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of difficulty urinating and statistics the number of participants who developed these symptoms
Number of participants who fell difficulty urinating at certain checkpoint of transplantation | 180 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of difficulty urinating and statistics the number of participants who developed these symptoms
Number of participants who fell difficulty urinating at certain checkpoint of transplantation | 360 days before transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of difficulty urinating and statistics the number of participants who developed these symptoms
Number of participants who fell lethargy at certain checkpoint of transplantation | 5 days before transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of lethargy and statistics the number of participants who developed these symptoms
Number of participants who fell lethargy at certain checkpoint of transplantation | 6 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of lethargy and statistics the number of participants who developed these symptoms
Number of participants who fell lethargy at certain checkpoint of transplantation | 30 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of lethargy and statistics the number of participants who developed these symptoms
Number of participants who fell lethargy at certain checkpoint of transplantation | 60 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of lethargy and statistics the number of participants who developed these symptoms
Number of participants who fell lethargy at certain checkpoint of transplantation | 100 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of lethargy and statistics the number of participants who developed these symptoms
Number of participants who fell lethargy at certain checkpoint of transplantation | 180 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of lethargy and statistics the number of participants who developed these symptoms
Number of participants who fell lethargy at certain checkpoint of transplantation | 360 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of lethargy and statistics the number of participants who developed these symptoms
Number of participants who fell dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia at certain checkpoint of transplantation | 5 days before transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia and statistics the number of participants who developed these symptoms
Number of participants who fell dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia at certain checkpoint of transplantation | 6 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia and statistics the number of participants who developed these symptoms
Number of participants who fell dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia at certain checkpoint of transplantation | 30 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia and statistics the number of participants who developed these symptoms
Number of participants who fell dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia at certain checkpoint of transplantation | 60 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia and statistics the number of participants who developed these symptoms
Number of participants who fell dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia at certain checkpoint of transplantation | 100 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia and statistics the number of participants who developed these symptoms
Number of participants who fell dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia at certain checkpoint of transplantation | 180 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia and statistics the number of participants who developed these symptoms
Number of participants who fell dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia at certain checkpoint of transplantation | 360 days after transplantation
  Use the Clinical Study Case Reports sheet to record whether each participant developed symptoms of dizziness, difficulty breathing, biliary colic, headache, stomachache, or anorexia and statistics the number of participants who developed these symptoms

IPD SHARING:
Plan to Share IPD: No